CLINICAL TRIAL: NCT00005405
Title: Parity and Serum Lipids in White and Hispanic Women
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4322; R03HL046168 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To analyze the relationships between parity (childbirth) or gravidity (pregnancy) and measures of lipids in groups of women from the Hispanic Health and Nutrition Examination Survey (Hispanic HANES) and the Framingham Heart Study.

DETAILED DESCRIPTION:
BACKGROUND:

The relationships between parity or gravidity and measures of lipids in groups of women from the Hispanic Health and Nutrition Examination Survey (Hispanic HANES) and the Framingham Heart Study offered insights into the health of an important minority group in the United States and provided clues regarding hormonal mechanisms in lipoprotein metabolism.

DESIGN NARRATIVE:

In the Framingham cohort, the relationships among gravidity, LDL-cholesterol, HDL-cholesterol and total cholesterol were prospectively studied. Each of these serum lipids was tested as a potential mediator of associations between gravidity and various cardiovascular endpoints. In the Hispanic HANES, the associations among parity, gravidity, and lipid levels were examined in cross-sectional data on women of a different ethnic background in whom birth rates tended to be high. Secondary analysis of these two datasets was conducted, carefully considering aspects of the study designs. Bivariate analyses generated mean lipid levels within parity or gravidity groups. HDL, LDL, and total cholesterol were then stratified both by parity and other variables (such as age and smoking status) so that interactions could be considered. Multivariate analyses were used to analyze the effect of parity on lipids and cardiovascular disease events while controlling for a variety of potentially confounding factors (such as body mass index, subscapular/triceps, skinfold ratio, education, income, cigarette smoking, alcohol consumption, oral contraceptive use, estrogen replacement therapy, menopausal status and type of menopause). Interactions were also considered in multivariate models.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09; Primary Completion 1993-09 (Actual); Study Completion 1993-09 (Actual)